CLINICAL TRIAL: NCT01026051
Title: A Phase 2, Open Label, Non-Randomized Study to Evaluate the Safety, Tolerability, Immune Response and Clinical Response of Multiple Doses of MKC1106-MT in Subjects With Advanced Melanoma
Brief Title: Safety, Immune and Tumor Response to a Multi-component Immune Based Therapy (MKC1106-MT) for Patients With Melanoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Financial/Business Reasons
Sponsor: Mannkind Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MKC1106-MT-002
Record Dates: First submitted 2009-12-03; First posted 2009-12-04 (Estimated); Last update posted 2012-05-15 (Estimated); Status verified 2012-05

CONDITIONS: Stage III Melanoma; Stage IV Melanoma
Keywords: Cancer Vaccine, Immunotherapy, Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: MKC1106-MT — Cancer Vaccine, Immunotherapy, Melanoma

SUMMARY:
The clinical trial is evaluating a multi-component active immunotherapy designed to stimulate an immune reaction to specific tumor associated antigens which are highly expressed on melanoma

DETAILED DESCRIPTION:
The multi-component active immunotherapy, MKC1106-MT, consists of 1 plasmid dose and 2 peptides doses designed to stimulate an immune reaction to two tumor associated antigens (Melan-A and tyrosinase). The plasmid component will be administered on Days 1, 4, 15 and 18 of each treatment cycle followed by administration of peptides on Days 29 and 32 of the treatment cycle. All components will be administered separately into non-diseased superficial inguinal lymph nodes under ultrasound guidance

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of regional or distant metastatic melanoma (stage IIIB, IIIC, or IV) confined to skin, subcutaneous tissue, or lymph nodes that is refractory to standard of care, or for which no curative standard therapy exists (Note: Subjects who are therapy-naïve will also be eligible.)
* Measurable disease by the Response Evaluation Criteria in Solid Tumours (RECIST) 1.1 criteria
* ECOG performance status of 0 or 1
* Life expectancy > or = 3 months
* 18 years of age or older at screening evaluation
* Subjects must be able to provide informed consent for participation in the clinical trial before any protocol-specific clinical trial procedure is performed
* Positive for HLA-A2 and, more precisely, for expression of A*0201 as assessed by DNA typing
* Tumor material from prior biopsy/surgical resection available for analysis of expression of melanoma specific antigens
* Adequate coagulation function as evidenced by prothrombin time (PT) and partial thromboplastin time (PTT) values within the normal range
* Adequate bone marrow reserve as evidenced by Absolute neutrophil count (ANC) > or = 1,000/mL; platelet count > or = 75,000/mL
* Subjects must have recovered to at least baseline or Grade 1 toxicity from the effects of any prior surgery, radiotherapy, or other therapies including but not limited to chemotherapy
* Women of childbearing potential as well as fertile men and their partners must agree to use an effective method of contraception or to abstain from sexual intercourse during the clinical trial and for 90 days following the last dose of the investigational drug.
* Subjects who have received local radiation therapy (less than one-fourth of bone marrow) are eligible.

Exclusion Criteria:

* Subjects with visceral metastasis (Note: Subjects with stable CNS metastasis or fully treated CNS metastatic disease [eg, radiation therapy] are eligible.)
* Active infection requiring treatment
* Systemic inflammatory disease requiring chronic maintenance or suppressive therapy
* Positive antibody test result for HIV, hepatitis B, or hepatitis C
* History of allogeneic transplant
* Medical, sociological, or psychological conditions that may compromise compliance or participation or that may interfere with the interpretation of the results
* History of receiving immunosuppressive drugs within 1 month before dosing
* Subjects who are lactating, pregnant, or planning to become pregnant within 3 months of completing treatment
* Subjects who received an investigational drug within the 4 weeks before dosing
* Prior systemic radiation therapy (more than one-fourth of bone marrow)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2010-10; Primary Completion 2011-09 (Actual); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
To evaluate the objective response, where response is defined as either complete response (CR), partial response (PR), or stable disease (SD) for 12 weeks or longer (CR, PR, and SD are defined according to RECIST 1.1 criteria) | 12 Months

SECONDARY OUTCOMES:
To assess clinical efficacy of MKC1106-MT in subjects with advanced melanoma measured at 6 months and 1 year by (1) time to progression, progression-free survival | 12 Months
To identify and characterize correlations between biological activity (immune response), target antigen expression and clinical efficacy. | 12 months
To further assess the safety profile and tolerability | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Chief Scientific Officer, Study Chair — Mannkind Corporation
Locations (4):
- United States (4):
  - The Angeles Clinic and Research Institute, Los Angeles, California
  - UCLA Medical Center, Los Angeles, California
  - Martin Memorial, Stuart, Florida
  - Nevada Cancer Institute, Las Vegas, Nevada